CLINICAL TRIAL: NCT03922594
Title: Surveillance of Zika-related Microcephaly in Sub-Saharan Africa and Asia
Status: Terminated | Type: Observational
Why Stopped: The disruptions due to the impact of the ongoing COVID-19 pandemic to the implementation of the study in each of the study sites, as well as to the coordination of the study at Institut Pasteur, prevented the completion of the study
Sponsor: Institut Pasteur (Industry)
Collaborators: Centre Pasteur du Cameroun (Other); Guangzhou Women and Children's Medical Center (Other); Institut Pasteur of Cote d'Ivoire (Other Government); Pasteur Institute, Ho Chi Minh City (Other Government); Tu Du Hospital (Other Government); Perinatal Society of Sri Lanka (Unknown); University of Colombo (Other); University of Lausanne (Other); University of Lausanne Hospitals (Other); The University of Hong Kong (Other); Ministry of Health of Sri Lanka (Unknown); Central Hospital Maternity (Unknown); Essos Hospital Center (Other); Guangzhou Baiyun Maternal and Child Health Hospital (Unknown); General Hospital of Yopougon-Attie (Unknown); General Hospital Abobo-Sud (Unknown); Castle Street Hospital for Women (Unknown); De Soyza Hospital for Women (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZIKA_2016-102
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-03

CONDITIONS: Microcephaly; Congenital Infection
MeSH Terms: conditions — Microcephaly | interventions — Diagnosis, Differential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cameroon: Live newborns with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns
  Interventions: Diagnostic Test: Differential diagnosis for infectious causes of microcephaly
- China: Fetuses or newborns (still-born, medical abortions or alive) with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns
  Interventions: Diagnostic Test: Differential diagnosis for infectious causes of microcephaly
- Ivory Coast: Live newborns with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex and severely disproportionate length or weight according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns
  Interventions: Diagnostic Test: Differential diagnosis for infectious causes of microcephaly
- Sri Lanka: Live newborns with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns
  Interventions: Diagnostic Test: Differential diagnosis for infectious causes of microcephaly
- Vietnam: Fetuses or newborns (still-born, medical abortions or alive) with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns
  Interventions: Diagnostic Test: Differential diagnosis for infectious causes of microcephaly

INTERVENTIONS:
Diagnostic Test: Differential diagnosis for infectious causes of microcephaly — Zika virus, cytomegalovirus, rubella, toxoplasmosis

SUMMARY:
This study will explore whether ZIKV is currently responsible for neurological complications, and particularly microcephaly, in Aedes-infested regions of Sub-Saharan Africa (SSA) and Asia. This will inform regional public health strategies, such as vaccination of women of child-bearing age. It will also demonstrate the public health impact of ZIKV infection and increase the understanding of other regional infectious (e.g. cytomegalovirus) causes of microcephaly.

DETAILED DESCRIPTION:
This study will last for 2 years, and will include only new cases of microcephaly.

Surveillance will take place in large maternities in urban areas (standard procedure)

* In each city, ~3000 live births per month will be monitored, so that on average one microcephaly will be diagnosed per month per city (i.e., 24 per city in 2 years)
* Microcephaly is defined as less than -3 standard deviation (SD), according to the INTERGROWTH standards by age and sex with abnormal ultrasound and/or clinical examination.

Data collection (study activity)

* A questionnaire with demographic, exposure and pregnancy details for all mothers Clinical exam and laboratory testing (standard procedure and study activity)
* Various biological samples (e.g. blood, placenta) will be collected from mothers and newborns/fetuses and tested for presence of ZIKV, and for other infectious (e.g. rubella, cytomegalovirus) causes of microcephaly
* Physical, neurological, hearing and visual examinations for all live births will be performed where possible.

Analysis and reporting (study activity)

o All results will be shared publically through conferences and peer-reviewed publications.

ELIGIBILITY:
Inclusion Criteria:

* All infants or fetuses with microcephaly, (defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex, detected during the mother's pregnancy, or at the end of the mother's pregnancy at one of the participating maternities)
* and with abnormal ultrasound and/or clinical examination findings for newborns.

Exclusion Criteria:

* Infants/fetuses with microcephaly whose mothers are under the age of 18 years,
* or inability or refusal of mothers/ guardians to give informed consent.

Ages: 0 Days to 2 Days | Sex: All
Age Groups: Child
Study Population: Fetuses or newborns (still-born, medical abortions [China and Vietnam only] or alive) with microcephaly defined as head circumference ≤-3SD according to INTERGROWTH standards for gestational age and sex with abnormal ultrasound and/or clinical examination findings for newborns.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of microcephaly (per 10,000 live births) | At birth
  Incidence of microcephaly (per 10,000 live births)
Proportion of microcephaly attributable to ZIKV | At birth
  Proportion of microcephaly attributable to Zika virus infection
Proportion of microcephaly linked to other infectious etiologies | At birth
  Proportion of microcephaly linked to other infectious etiologies (non-ZIKV)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Fontanet, Principal Investigator — Institut Pasteur
Locations (8):
- Cameroon (2):
  - Central Hospital Maternity, Yaoundé
  - Essos Hospital Centre Maternity, Yaoundé
- Guangzhou Women's and Children's Hospital, Guangzhou, China
- Côte d’Ivoire (2):
  - General Hospital Abobo-Sud, Abidjan
  - General Hospital of Yopougon-Attie, Abidjan
- Sri Lanka (2):
  - Castle Street Hospital for Women, Colombo
  - De Soyza Hospital for Women, Colombo
- Tu Du Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No